CLINICAL TRIAL: NCT00916448
Title: The Effects of Atazanavir-induced Hyperbilirubinemia on the Innate Immune Response During Human Endotoxemia. A Parallel Double Blind Placebo Controlled Pilot Study.
Brief Title: The Effects of Atazanavir-induced Hyperbilirubinemia During Human Endotoxemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ATV LPS study
Record Dates: First submitted 2009-06-05; First posted 2009-06-09 (Estimated); Last update posted 2015-08-14 (Estimated); Status verified 2015-07

CONDITIONS: Endotoxemia; Inflammation; Multi Organ Dysfunction Syndrome; Sepsis
Keywords: Endotoxin; Bilirubin; Inflammation; Sepsis; Multi organ dysfunction syndrome; Oxidative Stress; Heme oxygenase
MeSH Terms: conditions — Endotoxemia; Inflammation; Sepsis | interventions — Atazanavir Sulfate; endotoxin, Escherichia coli

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): placebo medication: 2 capsules taken twice daily for 4 consecutive days and thereafter infusion of 2 ng/kg E.coli endotoxin intravenously
  Interventions: Drug: E. coli endotoxin
- Atazanavir (Active Comparator): Atazanavir 150 mg, 2 capsules taken twice daily for 4 consecutive days and thereafter infusion of 2 ng/kg E.coli endotoxin intravenously
  Interventions: Drug: Atazanavir; Drug: E. coli endotoxin

INTERVENTIONS:
Drug: Atazanavir — capsules of 150 mg, 2 capsules, twice daily on 4 consecutive days
  Other Names: Reyataz
  Arms: Atazanavir
Drug: E. coli endotoxin — 2 ng/kg E. coli reference endotoxin 11:H 10:K negative intravenously

SUMMARY:
Excessive inflammation, production of free radicals and vascular injury are considered the main contributors to the development of organ dysfunction in patients with severe infections and sepsis. The endogenously produced unconjugated bilirubin is one of the most powerful anti-oxidants of the human body and the administration of bilirubin in animal experiments has been shown to protect from inflammation-induced death. However, bilirubin for human administration is not yet available. Therefore, we wish to exploit one of the side effects of atazanavir, a registered drug currently used as a protease inhibitor in HIV infected patients. Atazanavir inhibits the enzyme UPD glucuronosyl transferase enzyme (UGT1A1) and therefore increases endogenously produced bilirubin levels moderately. To study the effect of hyperbilirubinemia during inflammation we will apply the human endotoxemia model. The human endotoxemia model permits elucidation of key players in the immune response to a gram negative stimulus in vivo, therefore serving as a useful tool to investigate potential novel therapeutic strategies in a standardized setting. We hypothesize that atazanavir-induced hyperbilirubinemia has beneficial anti-inflammatory and vascular effects during human endotoxemia.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers

Exclusion Criteria:

* Use of any medication or anti-oxidant vitamin supplements.
* History of allergic reaction to atazanavir.
* Smoking.
* Previous spontaneous vagal collapse.
* History, signs or symptoms of cardiovascular disease.
* (Family) history of myocardial infarction or stroke under the age of 65 years.
* Cardiac conduction abnormalities on the ECG consisting of a 2nd degree atrioventricular block or a complex bundle branch block.
* Hypertension (defined as RR systolic > 160 or RR diastolic > 90).
* Hypotension (defined as RR systolic < 100 or RR diastolic < 50).
* Renal impairment (defined as plasma creatinin >120 μmol/l).
* Liver enzyme abnormalities or positive hepatitis serology.
* Subjects with a total bilirubin level above 15 μmol/L and a normal direct bilirubin level suggesting Gilbert Syndrome.
* Positive HIV serology or any other obvious disease associated with immune deficiency.
* Febrile illness in the week before the LPS challenge.
* Participation in a drug trial or donation of blood 3 months prior to the LPS challenge.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2009-05; Primary Completion 2010-03 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
The effect of atazanavir-induced hyperbilirubinemia on systemic activation of the innate immune response by measurement of various cytokines induced by a lipopolysaccharide (LPS) challenge. | before and at several time points until 24 hrs after endotoxin administration

SECONDARY OUTCOMES:
To determine if the attenuated vascular response to endothelium dependent vasodilators and vasoconstrictors during endotoxemia can be prevented by atazanavir-induced hyperbilirubinemia. | before and until 6 hours after endotoxin administration
To detect the effects of human endotoxemia on gastric perfusion measured by tonometry in the presence or absence of atazanavir-induced hyperbilirubinemia. | Before and at several time points up to 9 hours after endotoxin administration
To determine if atazanavir induced hyperbilirubinemia can attenuate subclinical renal damage (determined by several markers of acute kidney injury) known to occur during human endotoxemia. | Before and at several time points up to 24 hours after endotoxin administration
To determine the effect of atazanavir induced hyperbilirubinemia on heme oxygenase induction and activity during human endotoxemia. | before and at several time points up to 24 hours after endotoxin administration

CONTACTS AND LOCATIONS:
Overall Officials: Peter Pickkers, MD, PhD, Principal Investigator — Radboud University Nijmegen Medical Centre, The Netherlands
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Derived] Dorresteijn MJ, Dekker D, Zwaag J, Heemskerk S, Roelofs HMJ, Smits P, van der Hoeven JG, Wagener FADTG, Pickkers P. Atazanavir-induced unconjugated hyperbilirubinemia prevents vascular hyporeactivity during experimental human endotoxemia. Front Immunol. 2023 May 16;14:1176775. doi: 10.3389/fimmu.2023.1176775. eCollection 2023. PMID 37261364